CLINICAL TRIAL: NCT03459313
Title: Prevention of Injuries in Young Athletics (Track and Field) Athletes: Initiation of Life-long Sports Health Literacy - KLUB§ Athletics
Brief Title: Prevention of Injuries in Young Athletics (Track and Field) Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Swedish Athletics Association (Unknown)
Responsible Party: Principal Investigator, Jenny Jacobsson, PhD, Principal Investigator, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017/520-31
Record Dates: First submitted 2018-02-23; First posted 2018-03-08 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Sports Injury
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): The active group will be provided the intervention program, i.e. access to a website.
  Interventions: Other: Active group
- Control group (No Intervention): The control group will continue to train according to their routines and will get access to the website after 4 months.

INTERVENTIONS:
Other: Active group — For this study, the Frisk.Friidrott (Healthy.Athletics/Track&Field) website has been developed. The purpose of the website is to provide an easy-to-use tool that can assist coaches and parents involved in youth athletics with information how to structure training and recovery planning, provide guidance on possible injuries, and provide other information on health for youth athletes.
  Arms: Active group

SUMMARY:
The long-term purpose of an on-going participatory action research program "The KLUB-study" in Sweden, that involves scientists and representatives from all levels of athletics, is to develop a sustainable framework for safe athletics (track and field) training for child athletes born 2002-2006. The first part of the research program, a 1-year longitudinal study analysing training and injury data, was completed in November 2017. The present study sets out to evaluate a website that aims to support coaches and caregivers in their role as adult key stakeholders to foster young athletes to become adult athletes who possess the tools to maintain a healthy sporting lifestyle.

DETAILED DESCRIPTION:
The intervention will be implemented in youth athletics and evaluated in a randomised controlled trial (RCT). It will follow the consensus guidelines for studies in athletics and be reported according to the CONSORT checklist. The participating clubs will be randomly allocated into active and control group. The active group will be provided the intervention program, i.e. access to a website, aimed to support coaches, caregivers´ and athletes' and improve knowledge and health literacy to make more informed choices that promote health. The control group will continue to train according to their routines and will get access to the website after 4 months.

The participants will be assessed at three times, at the beginning of the study (T1), after four months (T2), at ten months (T3) and additional prospective data on training and injury will be collected during the first four months (T1b).

ELIGIBILITY:
Inclusion Criteria:

* belonging to a sports club and participate in organized training, athletics (track and field)
* born 2002 - 2006

Exclusion Criteria:

* not, on a regular basis, participating in athletics (track and field) training

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2018-03-18 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Injury incidence | four months
  The primary outcome measure will be time from study entry to the first reported injury event

SECONDARY OUTCOMES:
Health literacy | four and ten months
  Evaluate health literacy using Swedish versions of; The Japanese Communicative and Critical Health literacy scale (adults) and the Health Literacy for School-aged Children (HLSAC) instrument (youth athletes)

CONTACTS AND LOCATIONS:
Locations (1):
- Swedish Athletics, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobsson J, Timpka T, Ekberg J, Kowalski J, Nilsson S, Renstrom P. Design of a protocol for large-scale epidemiological studies in individual sports: the Swedish Athletics injury study. Br J Sports Med. 2010 Dec;44(15):1106-11. doi: 10.1136/bjsm.2009.067678. Epub 2010 May 19. PMID 20484318
- [Background] Jacobsson J, Bergin D, Timpka T, Nyce JM, Dahlstrom O. Injuries in youth track and field are perceived to have multiple-level causes that call for ecological (holistic-developmental) interventions: A national sporting community perceptions and experiences. Scand J Med Sci Sports. 2018 Jan;28(1):348-355. doi: 10.1111/sms.12929. Epub 2017 Aug 4. PMID 28605065
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893
- [Background] Timpka T, Alonso JM, Jacobsson J, Junge A, Branco P, Clarsen B, Kowalski J, Mountjoy M, Nilsson S, Pluim B, Renstrom P, Ronsen O, Steffen K, Edouard P. Injury and illness definitions and data collection procedures for use in epidemiological studies in Athletics (track and field): consensus statement. Br J Sports Med. 2014 Apr;48(7):483-90. doi: 10.1136/bjsports-2013-093241. PMID 24620036
- [Derived] Jacobsson J, Kowalski J, Timpka T, Hansson PO, Spreco A, Dahlstrom O. Universal prevention through a digital health platform reduces injury incidence in youth athletics (track and field): a cluster randomised controlled trial. Br J Sports Med. 2023 Mar;57(6):364-370. doi: 10.1136/bjsports-2021-105332. Epub 2022 Dec 23. PMID 36564148